CLINICAL TRIAL: NCT04575389
Title: the Association Between Serum Uric Acid Levels and the Risk of Metabolic Syndrome in Type 2 Diabetes Mellitus
Brief Title: Relation Between Serum Uric Acid and Metabolic Syndrome in Type 2 DM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Tarek Mahmoud Ahmed, doctor, Assiut University
Other Study IDs: metabolic risk factor
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum uric acid levels ,HBA1C , fasting plasma glucose ,lipid profile , creatinine level — diagnostic tests

SUMMARY:
This study will be undertaken to evaluate the association of serum uric acid (SUA) level with metabolic risk factors in patients with type 2 diabetes and their relation to eGFR status

DETAILED DESCRIPTION:
Metabolic syndrome (syndrome X, insulin resistance) is a multifactorial disease with multiple risk factors that arises from insulin resistance accompanying abnormal adipose deposition and function . It comprises a combination of risk factors for coronary heart disease, as well as for diabetes type 2 , fatty liver, and several cancers.

Sign and symptoms are ; Hypertension... Hyperglycemia.. Hypertriglyceridemia... Reduced high-density lipoprotein cholesterol (HDL-C).. Abdominal obesity... Chest pain or shortness of breath: Suggesting the rise of cardiovascular and other complications.. The prevalence of the metabolic syndrome is often more in the urban population of some developing countries than in its Western counterparts . The syndrome feeds into the spread of the diseases like type 2 diabetes, coronary diseases, stroke, and other disabilities. The present trend is not sustainable unless a magic cure is found (unlikely) or concerted global/governmental/societal efforts are made to change the lifestyle that is promoting it.

There has been a renewed interest in the association of uric acid with diabetes and its complications. Uric acid is a product of purine metabolism. Increased serum uric acid (SUA) level has been shown to be associated with hypertension(1) cardiovascular disease (CVD)(2) and chronic kidney disease(3) . Elevated SUA level was also associated with metabolic syndrome in both normal subjects as well as in patients with type 2 diabetes. And with type 2 diabetes mellitus(4) Higher SUA level independently predicted the incidence of type 2 diabetes in subjects who had abnormal fasting glucose levels (5) . It has been shown that SUA levels are higher in patients with prediabetic conditions and in patients with type 2 diabetes compared with the level in normal controls (6) . SUA level has been shown to be positively associated with all cause mortality risk, but cardiovascular mortality was associated with SUA level only among those with hyperglycemia (prediabetes and type 2 diabetes)(8) . Hyperuricemia has been found to be associated with risk factors of diabetes such as obesity and insulin resistance(9) . Uric acid has also been reported to be involved in the endothelial dysfunction by impairing nitric oxide production and causing inflammation(10) , These effects of uric acid likely account for its impact on CVD incidence(11) . In acute ischaemic stroke, the survivors with both lower (<4.7 mg/dL) and higher (>6.7 mg/dL) baseline SUA levels had poor outcomes after a 12 month follow up when compared with those who had SUA levels in the range of 4.7-6.7 mg/dL. This is suggestive of the protective nature of uric acid when it is within the optimal range.

SUA level was positively associated with increased incidence of cardiovascular diseases (CVD) in patients with abnormal eGFR (<90 mL/min/1.73 m2) . HbA1c was found to be inversely associated with hyperuricemia in patients with normal eGFR level (≥90 mL/min/1.73 m2). Incidence of metabolic syndrome did not show any relationship with SUA level. However, the incidence of hypertension, a component of metabolic syndrome, was significantly higher among patients with hyperuricemia. Waist circumference and serum triglycerides were higher, whereas serum high-density lipoprotein level was lower in patients with higher SUA level. (12) Serum urea and creatinine were elevated in hyperuricemic patients, suggesting impaired kidney function. Hyperuricemia is known to be associated with the decrease in kidney function (13) and because chronic kidney disease itself elevates SUA level,(14) it is difficult to interpret the causes of the elevated serum urea and creatinine in hyperuricemia. However, eGFR values were only slightly lower in hyperuricemic patients. Correlation analysis showed that both serum urea and creatinine levels were positively associated with SUA level.. This association was found to be significant in patients with normal eGFR levels as well. However, eGFR appears to be negatively associated with SUA level in patients with abnormal eGFR level. Decreased urine output leads to decreased excretion of uric acid, resulting in the elevated SUA level. Therefore, reduction in eGFR may increase SUA levels in these patients.

The importance of uric acid has been increasingly appreciated because of its association with the development of diabetes mellitus and related diseases. SUA level and susceptibility to hyperuricemic conditions depend on the factors such as gender, age and ethnicity. (15) With the increasing incidence of diabetes studying the impact of hyperuricemia in patients with diabetes is necessary.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patient

Exclusion Criteria:

1. patients with type 1 diabetes
2. gestational diabetes
3. patients with drug affecting uric acid levels
4. secondary diabetes

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient will be collected randomly from outpatient clinics of diabetic center of assiut univeristy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
the association of serum uric acid (SUA) level with metabolic risk factors in patients with type 2 diabetes | baseline
  the incidence of hypertension, a component of metabolic syndrome, is significantly higher among patients with hyperuricemia. Waist circumference and serum triglycerides are higher, whereas serum high-density lipoprotein level is lower in patients with higher SUA level.

REFERENCES:
- [Background] Bellows JG. Editorial: Continuing education in ophthalmology. Ann Ophthalmol. 1976 Jun;8(6):649. No abstract available. PMID 937945
- [Background] Fontelo P, Liu F. Finding translational science publications in MEDLINE/PubMed with translational science filters. Clin Transl Sci. 2011 Dec;4(6):455-9. doi: 10.1111/j.1752-8062.2011.00320.x. Epub 2011 Nov 7. PMID 22212228
- [Background] Pozas E, Pascual M, Nguyen Ba-Charvet KT, Guijarro P, Sotelo C, Chedotal A, Del Rio JA, Soriano E. Age-dependent effects of secreted Semaphorins 3A, 3F, and 3E on developing hippocampal axons: in vitro effects and phenotype of Semaphorin 3A (-/-) mice. Mol Cell Neurosci. 2001 Jul;18(1):26-43. doi: 10.1006/mcne.2001.0999. PMID 11461151
- [Background] Wang XR, Robinson KM, Carter-Harris L. Prevalence of chronic illnesses and characteristics of chronically ill informal caregivers of persons with dementia. Age Ageing. 2014 Jan;43(1):137-41. doi: 10.1093/ageing/aft142. Epub 2013 Sep 26. PMID 24072413
- [Background] Turner AJ, Hick PE. Inhibition of aldehyde reductase by acidic metabolites of the biogenic amines. Biochem Pharmacol. 1975 Sep 15;24(18):1731-3. doi: 10.1016/0006-2952(75)90016-7. No abstract available.
- [Background] Kunkler I, Jack W, Prescott R, Williams L, King C. Postoperative breast irradiation: new trials needed in older patients. J Clin Oncol. 2003 May 1;21(9):1893; author reply 1893-4. doi: 10.1200/jco.2003.99.239. No abstract available. PMID 12721273
- [Background] Woods DJ. Conceptualizing depression and its treatment: comparison of psychoanalytic and behavioral approaches. Psychol Rep. 1975 Dec;37(3 PT 2):1271-8. doi: 10.2466/pr0.1975.37.3f.1271. No abstract available. PMID 1823
- [Background] Dupuy B, Mounier J, Blanquet P. [Some comments on the biological properties of calcitonin: an eventual new therapeutic utilization (author's transl)]. Ann Endocrinol (Paris). 1977 Jul-Aug;38(4):323-6. French. PMID 561566
- [Background] Fritsch P, Honigsmann H, Jaschke E, Wolff K. [Photochemotherapy of psoriasis: increasing its effectiveness with an oral aromatic retinoid (clinical results in 134 patients) (author's transl)]. Dtsch Med Wochenschr. 1978 Nov 3;103(44):1731-6. doi: 10.1055/s-0028-1129333. German. PMID 361362
- [Background] Bundgaard H. Polymerization of penicillins: kinetics and mechanism of di- and polymerization of ampicillin in aqueous solution. Acta Pharm Suec. 1976;13(1):9-26. No abstract available. PMID 3942